CLINICAL TRIAL: NCT06678165
Title: A Pilot Study on the Safety and Efficacy of YOLT-204 for Transfusion-Dependent Beta-Thalassemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOLT-204-IIT
Record Dates: First submitted 2024-10-31; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Transfusion Dependent Beta Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The intervention group will receive YOLT-204 on day0 (Experimental)
  Interventions: Drug: YOLT-204

INTERVENTIONS:
Drug: YOLT-204 — The intervention group will receive YOLT-204 on day0

SUMMARY:
This study is a single-arm, open-label, dose-escalation trial, planning to enroll 3-9 patients with transfusion-dependent β-thalassemia, aimed at assessing the safety and tolerability of a single-dose of YOLT-204 in patients with transfusion-dependent β-thalassemia; to preliminarily evaluate the impact of a single -dose of YOLT-204 on the levels of fetal hemoglobin in the plasma

ELIGIBILITY:
Inclusion Criteria：

1. Age between 18 to 35 years, gender not limited.
2. The patient has fully understood this study and voluntarily signed an informed consent form.
3. Clinically diagnosed as a patient with transfusion-dependent β-thalassemia, excluding the genotype: β0β0.
4. Karnofsky Performance Status (KPS) score of at least 70.
5. Obtain detailed medical records of red blood cell transfusions within 2 years prior to the patient signing the informed consent form, including the volume or units of transfusion and the levels of red blood cells and hemoglobin before and after transfusion.
6. No severe hematopoietic dysfunction, with heart, lung, liver, and kidney functions essentially normal.
7. Coagulation function: International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) both ≤1.5×ULN (Upper Limit of Normal).
8. Renal function: Creatinine ≤1.5×ULN, or when creatinine >1.5×ULN, the creatinine clearance is >50ml/min (calculated according to the Cockcroft-Gault formula).
9. Liver function: Alanine Aminotransferase (ALT) ≤3×ULN and Aspartate Aminotransferase (AST) ≤3×ULN; Direct Bilirubin ≤2.5×ULN.
10. Cardiac function: Left Ventricular Ejection Fraction (LVEF) ≥50%.
11. Good compliance, willing to adhere to visit schedules, trial plans, laboratory tests, and other trial steps.
12. Willing to participate in long-term follow-up studies.

Exclusion Criteria:

1. History of multiple drug allergies or a history of allergic reactions to oligonucleotides or lipid nanoparticles (LNPs).
2. Diagnosed with compound alpha-thalassemia.
3. Clinically significant active bacterial, viral, fungal, or parasitic infections at the time of screening, as judged by the investigator.
4. White blood cell count (WBC) <3×10^9/L and/or platelet count <100×10^9/L not due to hypersplenism, as judged by the investigator.
5. Uncorrected bleeding disorders.
6. Received treatment with erythropoietin (EPO) within the three months prior to enrollment.
7. Severe iron overload, with serum ferritin levels ≥5000 ng/ml.
8. Positive for hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus, antibodies to human immunodeficiency virus (HIV), or specific antibodies to Treponema pallidum (syphilis).
9. History of hematopoietic stem cell transplantation, gene therapy, or gene editing therapy.
10. Participation in another clinical study and use of investigational drugs within 3 months prior to starting the study drug.
11. History or current presence of malignant tumors or myeloproliferative diseases or immunodeficiency diseases.
12. Presence of severe mental illness that prevents cooperation with treatment; significant pulmonary arterial hypertension requiring medical intervention; recent malaria; a history of hematological tumors in immediate family members.
13. Any past or current disease, treatment, or laboratory abnormality that may interfere with the study results, affect the patient's full participation in the study, or that the investigator deems unsuitable for participation in this clinical study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 52 weeks after dose
  Number of Participants with Treatment-Emergent Adverse Events
Laboratory Test Findings | 52 weeks after dose
  Number of Participants with Clinically Significant Clinical Laboratory Test Findings
Safety Measurements | 52 weeks after dose
  Number of Participants with Clinically Significant Safety Measurements
3 months of sustained transfusion reduction | 4 months after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 3 months of sustained transfusion reduction (sustained TR3) is obtained.
3 months of transfusion independence | 4 months after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 3 months of transfusion independence (sustained TI3) is obtained.

SECONDARY OUTCOMES:
6 months of sustained transfusion reduction | 7 months after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 6 months of sustained transfusion reduction (sustained TR6) is obtained.
6 months of transfusion independence | 7 months after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 6 months of transfusion independence (sustained TI6) is obtained.
The proportion of alleles with intended modifications | 52 weeks after dose
  The proportion of alleles with intended modifications in peripheral blood leukocytes and bone marrow cells over time.
Fetal hemoglobin concentration | 52 weeks after dose
  The change in fetal hemoglobin concentration over time after YOLT-204 infusion
Total hemoglobin concentration | 52 weeks after dose
  The change in total hemoglobin concentration over time after YOLT-204 infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China